CLINICAL TRIAL: NCT01524185
Title: FamilyLive Feasibility and Effectiveness Study
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: There were not enough eligible families and trained clinicians to conduct RCT.
Sponsor: Hugo W. Moser Research Institute at Kennedy Krieger, Inc. (Other)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Harolyn M.E.Belcher, M.D., Director of Research, Family Center at Kennedy Krieger Institute, Hugo W. Moser Research Institute at Kennedy Krieger, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NA_00022038
Record Dates: First submitted 2012-01-30; First posted 2012-02-01 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Mood Lability; PTSD; Anxiety
Keywords: childhood trauma; intergenerational trauma; child neglect; child maltreatment; mental health
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Anxiety Disorders; Historical Trauma; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FamilyLive (Experimental): Multi-therapist group intervention for families with a history of intergenerational neglect and trauma exposure
  Interventions: Behavioral: FamilyLive
- Standard Mental Health Treatment (Active Comparator): Standard trauma-informed mental health treatment
  Interventions: Behavioral: Standard Mental Health Treatment

INTERVENTIONS:
Behavioral: FamilyLive — Multi-therapist family mental health treatment for families with a history of intergenerational neglect and trauma
  Other Names: FL
  Arms: FamilyLive
Behavioral: Standard Mental Health Treatment — Standard trauma-informed mental health treatment
  Other Names: SMHC
  Arms: Standard Mental Health Treatment

SUMMARY:
Children who have been exposed to trauma (defined as physical, sexual or emotional abuse, neglect, exposure to life threatening events, domestic and community violence, parental mental health disorders, substance abuse, and/or incarceration may also have parents who have experienced trauma. Often, unresolved intergenerational trauma makes treatment of children with trauma and its sequelae, including Post Traumatic Stress Disorder, attachment disorders and dysregulation characterized by emotional lability, hyperarousal, and sleep and attention disturbances, difficult to manage. FamilyLive (FL) is a promising treatment approach developed by clinicians at the Kennedy Krieger Family Center (KKFC) over 10 years ago to address the unique needs of families with unresolved and untreated histories of neglect and disrupted attachment who need support to build skills for managing their children's responses and behaviors. FL uses a team approach with a therapist in the room with the family and call-in observations and clinical suggests from a clinician behind a one-way mirror. Through the call-in process the treatment team provides validation, acknowledgement, support and multiple perspectives for the family's experiences. The FL approach works with families to improve parental self-care, stress management, emotional regulation and self-awareness.

Despite its clinical use at the KKFC, the effectiveness of the FL intervention not been systematically evaluated using a randomized design. The proposed preliminary study will use a randomized design to evaluate the feasibility of conducting a larger randomized trial of FL compared to other standard mental health care treatments (SMHC) at the KKFC. We hypothesize that it will be feasible to recruit sufficient numbers of clients for and conduct a randomized controlled trial of FL on a cohort of children exposed to neglect and trauma. We also hypothesize that FL participants will evidence greater reductions in heart rate variability, behavior problems, trauma symptoms, and improvements in functioning compared to participants in the SMHC.

DETAILED DESCRIPTION:
Children who have been exposed to neglect often have parents who experienced their own childhood neglect and/or trauma (defined as childhood physical, sexual or emotional abuse, exposure to life threatening events, domestic and/or community violence, parental mental health disorders, substance abuse, and/or incarceration). These parental experiences of neglect and trauma during childhood are associated with disengaged and ineffective parenting behaviors and disrupted attachment processes between the parent and their own child. Disrupted attachment can result in the child exhibiting physiological dysregulation and behavior problems, which pose barriers to the child's academic and social success/development. Often, unresolved intergenerational trauma makes treatment of children with trauma and its sequelae, including Posttraumatic Stress Disorder, attachment disorders and dysregulation characterized by emotional lability, hyperarousal, and sleep and attention disturbances, difficult to manage.

FamilyLive (FL) is a promising treatment approach developed by clinicians at the Kennedy Krieger Family Center (Family Center) over 10 years ago to address the unique needs of families with unresolved and untreated histories of neglect and disrupted attachment who need support to build skills for managing their children's responses and behaviors. FL uses a team approach with a therapist in the room with the family and call-in observations and clinical suggests from a clinician behind a one-way mirror. Through the call-in process the treatment team provides validation, acknowledgement, support and multiple perspectives for the family's experiences. The FL approach works with families to improve parental self-care, stress management, emotional regulation and self-awareness. Despite its clinical use at the Family Center, the effectiveness of FL has never been systematically evaluated using a randomized design.

This study will systematically evaluate the feasibility of conducting a randomized clinical trial of FL versus standard mental health care at the Family Center for children with a history of neglect and their caregivers who also have a history of childhood neglect, with or without trauma. Caregivers are defined as any adult who assumes primary responsibility for the child's daily care in the home environment, and may include a biological parent, adoptive parent, grandparent, aunt/uncle, sibling who has reached the age of majority who is the primary caretaker of the child client, etc. Evaluation methods include standardized instruments and EKG administered at baseline, 3, 6, and 12 months.

Study Objectives:

Primary objective: To examine the feasibility of recruiting and conducting the proposed intervention and evaluation procedures on a cohort of children exposed to neglect and their caregivers using a randomized design.

Secondary objective: Examine the effects of FL on heart rate variability, behavior, post traumatic stress disorder symptoms, and functioning.

Tertiary objective: To examine differences in treatment outcomes (trauma symptoms, behavior problems, child functioning, parent behavior, etc.) between clients who receive FamilyLive and clients who receive SMHC at the Family Center.

ELIGIBILITY:
Inclusion criteria:

* Children, ages 5-17 years 11 months,
* enrolled in treatment at KKFC and each child's primary caregiver will be invited to participate if the child continues to exhibit behavior dysregulation (CBCL of > 60) and/ or attachment difficulties following 3 months of SMHC at the KKFC and if parents have a history of neglect (with or without trauma).

Exclusion criteria:

* Children with cardiac arrhythmias, endocrine disorders associated with heart rate irregularities or who are not able to cooperate or understand study procedures will be excluded.
* Non-English speaking children or hearing impaired will be excluded.
* Children in foster care.

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-02; Primary Completion 2016-01-08 (Actual); Study Completion 2016-01-08 (Actual)

PRIMARY OUTCOMES:
To examine the feasibility of recruiting and conducting the proposed intervention and evaluation procedures on a cohort of children exposed to neglect and their caregivers using a randomized design. | 4 years

SECONDARY OUTCOMES:
Examine the effects of FL on heart rate variability, behavior, post traumatic stress disorder symptoms, and functioning | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Kennedy Krieger Institute, Baltimore, Maryland, United States